CLINICAL TRIAL: NCT02269943
Title: A Phase 2, Multicenter, International, Single Arm Study To Assess The Safety And Efficacy Of Single Agent Cc-486 (Oral Azacitidine) In Previously Treated Subjects With Locally Advanced Or Metastatic Nasopharyngeal Carcinoma
Brief Title: Safety and Efficacy of CC-486 in Previously Treated Patients With Locally Advanced or Metastatic Nasopharyngeal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-486-NPC-001; 2014-001745-25 (EudraCT Number)
Expanded Access: NCT03723135 (Approved for marketing)
Record Dates: First submitted 2014-10-17; First posted 2014-10-21 (Estimated); Results first posted 2018-06-01 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-11

CONDITIONS: Nasopharyngeal Neoplasms
Keywords: Metastatic nasopharyngeal carcinoma; oral azacitidine; oral AZA; CC-486; metastatic; recurrent; nasopharyngeal carcinoma; nasal; solid tumors; locally advanced; rare head and neck cancer; nasopharynx; single chemotherapy agent; Epstein-Barr Virus (EBV) + nasopharyngeal carcinoma; EBV-DN; Celgene; Sponsor-study; oral chemotherapy; phase 2; oral Vidaza; EBV promoter methylation; hypomethylation; tumor infiltrating lymphocytes (TILs); EBV gene expression; neoplasms
MeSH Terms: conditions — Nasopharyngeal Neoplasms; Nasopharyngeal Carcinoma; Neoplasm Metastasis; Recurrence; Head and Neck Neoplasms; Epstein-Barr Virus Infections; Neoplasms | interventions — cc-486; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CC-486 (Experimental): CC-486 will be administered orally every day on Days 1-14 of a 21 day cycle at a dose of 300 mg. The first 6 participants of Asian-Pacific ethnicity will receive a starting dose of 200 mg. If there are no safety concerns, the 300 mg dose will be administered to all subsequent participants of Asian-Pacific ethnicity.
  Interventions: Drug: CC-486

INTERVENTIONS:
Drug: CC-486
  Other Names: oral azacitidine

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of CC-486 in previously treated patients with locally advanced or metastatic nasopharyngeal carcinoma having failed one to two previous regimens, including platinum-based chemotherapy. Participants will be enrolled according to a Simon two-stage design; if the predefined activity is met (>4 responses [complete response; partial response {CR/PR}] out of the first 17 evaluable participants based on independent radiological assessment), then the study will continue to enroll an additional 34 participants. If 4 or less responses out of 17 are observed, then the study enrollment will be stopped.

ELIGIBILITY:
Inclusion Criteria:

* Age = or > 18 years Histological or cytological diagnosis of undifferentiated or poorly differentiated nasopharyngeal carcinoma that is locally advanced or metastatic.
* Disease progression either clinically or radiographically after 1-2 previous regimens.
* Patient has received a platinum containing regimen. Eastern Cooperative Oncology Group (ECOG) performance status 0-2. Radiographically-documented measureable disease.
* Adequate organ and bone marrow functions.
* Willingness to follow pregnancy precautions.

Exclusion Criteria:

* History of, or current brain metastasis. Any other malignancy within 5 years prior to randomization with the exception of adequately treated in situ carcinoma of the cervix, uteri, or non-melanomatous skin cancer (all treatment of which should have been completed 6 months prior to enrollment), in situ squamous cell carcinoma of the breast, or incidental prostate cancer.
* Previous treatment with azacitidine (any formulation), decitabine, any other hypomethylating agent.
* History of gastrointestinal disorder or defect. Impaired ability to swallow oral medication. Persistent diarrhea or malabsorption.
* Active cardiac disease and human immunodeficiency virus (HIV) infection
* Active bleeding; pathological condition that carries a high risk of bleeding; risk of pseudoaneurysm of the internal carotid artery and carotid blowout syndrome.
* Major surgery within 14 days prior to starting Investigational Product or has not recovered from major side effects.
* Another investigational therapy within 28 days or 5 half lives of randomization/enrollment, whichever is shorter.
* Patient has not recovered from the acute toxic effects of prior anticancer therapy, radiation, or major surgery/significant trauma.
* Radiotherapy < or = 4 weeks or limited field radiation for palliation < or = 2 weeks prior to starting with the investigational product.
* Pregnancy/Breast feeding
* Any condition that places the patient at unacceptable risk if he/she were to participate in the study or that confounds the ability to interpret data from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-02-13 (Actual); Primary Completion 2017-04-20 (Actual); Study Completion 2017-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abderahim (Rahim) Fandi, MD, PhD, Study Director — Celgene
Locations (25):
- United States (5):
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Columbia Comprehensive Cancer Care Clinic, Jefferson City, Missouri
  - Levine Cancer Institute, Charlotte, North Carolina
- Canada (2):
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - McGill University, Montreal, Quebec
- France (3):
  - Institut Hospitalier Franco-Britannique, Levallois-Perret
  - Institut Curie, Paris
  - Institut Gustave Roussy, Villejuif
- Greece (2):
  - University General Hospital of Heraklion, Heraklion
  - Thermi Clinic, Thessaloniki
- Istituto Nazionale Dei Tumori, Milan, Italy
- Singapore (3):
  - National Cancer Center, Singapore
  - Singapore Oncology Consultants, Singapore
  - Johns Hopkins Singapore International Medical Centre, Singapore
- Spain (3):
  - Instituto Catalan de Oncologia-Hospital Duran, Barcelona
  - Hospital Universitario Madrid Sanchinarro, Madrid
  - Hospital Universitario de Salamanca, Salamanca
- Taiwan (3):
  - Chang Gung Medical Foundation, Kaohsiung Memorial Hospital, Niao-Sung Hsiang Kaohsiung County
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
- Tunisia (3):
  - Hopital Abderrahman Mami de Pneumo-Phtisiologie de l'Ariana, Aryanah
  - Institut Salah Azaiez, Bab Saadoun
  - Hospital Habib Bourguiba, Sfax

REFERENCES:
- [Derived] Von Hoff DD, Rasco DW, Heath EI, Munster PN, Schellens JHM, Isambert N, Le Tourneau C, O'Neil B, Mathijssen RHJ, Lopez-Martin JA, Edenfield WJ, Martin M, LoRusso PM, Bray GL, DiMartino J, Nguyen A, Liu K, Laille E, Bendell JC. Phase I Study of CC-486 Alone and in Combination with Carboplatin or nab-Paclitaxel in Patients with Relapsed or Refractory Solid Tumors. Clin Cancer Res. 2018 Sep 1;24(17):4072-4080. doi: 10.1158/1078-0432.CCR-17-3716. Epub 2018 May 15. PMID 29764853

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter study with 17 sites from the United States, Canada, France. Greece, Italy, Spain, Taiwan, Singapore and Tunisia.
Pre-assignment Details: Participants were enrolled according to a Simon 2-stage design. The first 6 participants of Asian-Pacific Island ethnicity received 200 mg/day CC-486 on days 1-14 of each 21-day cycle to monitor safety and tolerability; if there were no safety concerns, subsequent participants of Asian-Pacific Island ethnicity would receive the 300 mg daily dose
Groups:
- CC-486 200 mg: Asian-Pacific island participants received CC-486 200 mg tablets by mouth (PO) on days 1-14 of each 21-day cycle until radiologic disease progression, unacceptable toxicity, adverse event, a new anticancer therapy is begun, withdrawal of consent, subject refusal, physician decision, or death. If well tolerated, and there were no safety concerns, subsequent participants of Asian-Pacific Island ethnicity were administered CC-486 300-mg PO daily for 14 days of a 21-day cycle.
- CC-486 300 mg: Participants received CC-486 300 mg tablets by mouth on days 1-14 of each 21-day cycle until radiologic disease progression, unacceptable toxicity, adverse event (AE), a new anticancer therapy is begun, withdrawal of consent, subject refusal, physician decision, or death.
Period: Treatment Period
Arm/Group | CC-486 200 mg | CC-486 300 mg
Started | 6 | 30
Investigational Product (IP) Stopped (IP stopped due to disease progression, consent withdrawal, AE, discontinued at physician's decision) | 6 | 30
Completed | 0 (Not applicable according to the study design) | 0 (Not applicable according to the study design)
Not Completed | 6 | 30
Not completed — Death | 0 | 1
Not completed — Adverse Event | 1 | 10
Not completed — Progressive Disease | 5 | 17
Not completed — Symptomatic Deterioration | 0 | 2
Period: Follow-Up Survival Period
Arm/Group | CC-486 200 mg | CC-486 300 mg
Started | 5 | 26
Completed | 0 (Not applicable according to the study design.) | 0 (Not applicable according to the study design.)
Not Completed | 5 | 26
Not completed — Death | 3 | 16
Not completed — Lost to Follow-up | 0 | 2
Not completed — Alive | 2 | 8

BASELINE CHARACTERISTICS:
Population: Enrolled Population: The Enrolled Population included all participants who were enrolled to the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | CC-486 200 mg | CC-486 300 mg | Total
Number analyzed (Participants) | 6 | 30 | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.2 (11.70) | 52.2 (11.60) | 52.4 (11.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 4 | 25 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 6 | 7 | 13
  White | 0 | 23 | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 0 | 0 | 0
  Non-Hispanic or Latino | 6 | 30 | 36
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG performance status is used by doctors and researchers to assess how a subject's disease is progressing, assess how the disease affects the daily living activities of the subject and determine appropriate treatment and prognosis. 0 = Fully Active (Most Favorable Activity); 1 = Restricted activity but ambulatory; 2 = Ambulatory but unable to carry out work activities; 3 = Limited Self-Care; 4 = Completely Disabled, No self-care (Least Favorable Activity)
  Participants
    0 = Fully Active | 4 | 11 | 15
    1 = Restrictive but ambulatory | 2 | 18 | 20
    2 = Ambulatory but unable to work | 0 | 1 | 1
    3 = Limited Self-Care | 0 | 0 | 0
Time From Initial Diagnosis to First Dose [Mean (Standard Deviation); unit: years] | 3.60 (3.204) | 3.86 (3.358) | 3.81 (3.287)
Nasopharyngeal Cancer (NPC) Diagnosis Types [Count of Participants; unit: Participants] — The 3 types of NPC, based on how the cancer cells look under the microscope include:
  1. Undifferentiated Nasopharyngeal Carcinoma
  2. Poorly Differentiated Nasopharyngeal Carcinoma
  3. Other
  Participants
    Undifferentiated Nasopharyngeal Carcinoma | 2 | 21 | 23
    Poorly Differentiated Nasopharyngeal Carcinoma | 2 | 9 | 11
    Other | 2 | 0 | 2
Participants with Prior Anti-Cancer Therapies [Count of Participants; unit: Participants] — Population: The Safety Population included all participants who received at least
  1 dose of investigational product (IP)
  Participants | 6 | 29 | 35

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved a Complete or Partial Response According to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) Based on an Independent Radiology Assessment (IRA)
Description: Overall response rate was defined as the combined incidence of Complete Response (CR) or Partial Response (PR), confirmed no less than 4 weeks after the criteria for response were first met, based on independent radiology assessment according to RECIST 1.1 criteria.
  Complete response was defined as the disappearance of all target lesions and non-target lesions; Partial response is at least a 30% decrease from baseline in the sum of diameters of target lesions with no progression of non-target lesions and no new lesions or disappearance of target lesions with persistence of one or more non-target lesions from baseline.
Time Frame: Tumor response was assessed every (Q) 6 weeks for the first 3 evaluations then Q 9 weeks until disease progression as of the cut-off date of 08 August 2017; the median duration of treatment was 257 days for the 200 mg dose and 114.5 days for 300 mg dose
Population: The Efficacy Evaluable Population included all enrolled participants who met eligibility criteria and either received 2 cycles of CC-486 at any dose and discontinued treatment for progressive disease or received 4 cycles of CC-486 and had a baseline and at least 2 post-screening tumor assessments.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | CC-486 200 mg | CC-486 300 mg
Number analyzed (Participants) | 5 | 20
percentage of participants | 0 [NA to NA] — Confidence interval could not be calculated because there were no participants who had a response. | 15.0 [4.2 to 34.4]

2. Primary Outcome: Kaplan Meier Estimate of Progression-Free Survival (PFS) Based on an Independent Radiology Assessment According to RECIST 1.1 Criteria
Description: PFS was defined as the time from the date of start of the study treatment to the date of disease progression or death (any cause) on or prior to the data cut-off date for the statistical analysis, whichever occurred earlier, based on an independent radiology assessment of response using RECIST v1.1 criteria. Progressive disease was defined as at least a 20% increase in the sum of diameters of target or non-target lesions from nadir or appearance of a new lesion.
Time Frame: From Day 1 of documented disease progression; up to data cut off date of 08 August 2017; median follow-up time for censored participants was 12.3 months
Population: as for outcome 1
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | CC-486 200 mg | CC-486 300 mg
Number analyzed (Participants) | 5 | 20
months | 6.2 [1.4 to NA] — NA = Upper limit of the confidence interval (CI) for PFS could not be calculated because the upper limit was not reached due to limited number of events. | 4.4 [1.6 to 7.3]

3. Secondary Outcome: Kaplan Meier Estimate of Overall Survival
Description: Overall survival was the time from the first dose of study drug to patient death from any cause. Participants who did not die were censored at the last known time the patient was alive date or the clinical data cutoff date, whichever was earlier.
Time Frame: From Day 1 of study treatment to the first date of progressive disease or death; up to data cut-off date of 08 August 2017; overall median follow-up time for censored participants was 20.4 months
Population: as for outcome 1
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | CC-486 200 mg | CC-486 300 mg
Number analyzed (Participants) | 5 | 20
months | 18.0 [15.9 to NA] — NA = the CI for overall survival could not be calculated because the upper limit was not reached due to limited number of events. | NA [12.5 to NA] — NA = The median and upper limit of the CI for overall survival could not be calculated because the median or upper limit was not reached due to limited number of events.

4. Secondary Outcome: Percentage of Participants With Stable Disease for ≥ 16 Weeks From the Date of the First Treatment, or CR or PR According to RECIST 1.1 Criteria and Based on an Independent Radiology Assessment
Description: Disease Control Rate (DCR) was defined as the percentage of participants with a CR, PR, confirmed ≥ 4 weeks after the criteria for response were first met, or stable disease for ≥ 16 weeks from the first treatment, based on independent radiology assessment using RECIST 1.1 criteria. A complete response was defined as the disappearance of all target lesions and non-target lesions; a partial response is at least a 30% decrease from baseline in the sum of diameters of target lesions with no progression of non-target lesions and no new lesions or disappearance of target lesions with persistence of one or more non-target lesions from baseline. Stable disease is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase of lesions to qualify for progressive disease
Time Frame: Tumor response was assessed every 6 weeks for the first 3 evaluations then every 9 weeks until disease progression. As of the cut-off date of 08 August 2017 the median duration of treatment was 257 days for the 200 mg dose and 114.5 days for 300 mg dose
Population: Efficacy Evaluable Population = enrolled participants who met eligibility criteria and either received 2 cycles of IP at any dose and discontinued treatment for progressive disease or received 4 cycles of IP and had at least 2 post-screening tumor exams.
Measure: Median (90% Confidence Interval); unit: percentage of participants
Arm/Group | CC-486 200 mg | CC-486 300 mg
Number analyzed (Participants) | 5 | 20
percentage of participants | 60.0 [18.9 to 92.4] | 50.0 [30.2 to 69.8]

5. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: Treatment-emergent adverse events (TEAEs) were defined as any adverse event (AE) or serious adverse event (SAE) that occurred or worsened on or after the day of the first dose of the investigational product (IP) through 28 days after the last dose of IP. In addition, any SAE with an onset date more than 28 day after the last dose of IP that was assessed by the investigator as related to IP was considered a TEAE. The severity of AEs was graded based on National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE), Version 4.0 and based on the following scale: Grade 1 = Mild Grade 2 = Moderate Grade 3 = Severe Grade 4 = Life threatening Grade 5 = Death.
Time Frame: From date of first dose of study treatment to 28 days after last dose of study treatment; up to final data cut-off date of 08 August 2017; median treatment duration was 257 days for CC-486 200 mg and 114.5 days for CC-486 300 mg
Population: The Safety Population included all participants who received at least 1 dose of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | CC-486 200 mg | CC-486 300 mg
Number analyzed (Participants) | 6 | 30
Participants
  Any TEAE | 6 | 30
  Any TEAE Related to IP | 6 | 28
  Any Serious TEAE | 4 | 12
  Any Serious TEAE Related to IP | 3 | 7
  Any CTCAE Grade 3 or 4 TEAE | 6 | 20
  Any CTCAE Grade 3 or 4 TEAE Related to IP | 6 | 16
  Any TEAE Leading to Death | 1 | 1
  Any TEAE Leading to Dose Reduction | 5 | 9
  Any TEAE Leading to Drug Interruption | 4 | 9
  Any TEAE Leading to IP Discontinuation | 1 | 10

6. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration Of CC-486 (AUC-t)
Description: Area under the plasma concentration-time curve from Time 0 to the time of the last quantifiable concentration, calculated by linear trapezoidal method when concentrations are increasing and the logarithmic trapezoidal method when concentrations are decreasing.
Time Frame: Blood samples for oral azacitidine PK assessment were collected prior to each dose (pre-dose) and over the 8-hour period following each dose (0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, and 8 hours post-dose or similar schedule).
Population: The PK population includes participants with evaluable CC-486 plasma PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | CC-486 200 mg | CC-486 300 mg
Number analyzed (Participants) | 6 | 7
ng*h/mL
  Cycle 1 Day 1: number analyzed (Participants) | 4 | 6
  Cycle 1 Day 1 | 390.0 (58.8) | 351.7 (87.5)
  Cycle 1 Day 14: number analyzed (Participants) | 5 | 3
  Cycle 1 Day 14 | 130.3 (995.5) | 461.3 (104.2)

7. Secondary Outcome: Area Under the Plasma Concentration -Time Curve From 0 Extrapolated to Infinity (AUC-inf, AUC0-∞) Of CC-486
Description: Area under the plasma concentration-time curve from Time 0 extrapolated to infinity, calculated as [AUCt + Ct/ λz]. Ct is the last quantifiable concentration. No AUC extrapolation was performed with unreliable λz. If AUC %Extrap was ≥25%, AUC inf was not reported.
Time Frame: as for outcome 6
Population: The PK population includes participants with evaluable CC-486 plasma PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | CC-486 200 mg | CC-486 300 mg
Number analyzed (Participants) | 6 | 7
ng*h/mL
  Cycle 1 Day 1: number analyzed (Participants) | 4 | 6
  Cycle 1 Day 1 | 392.5 (58.3) | 354.9 (87.1)
  Cycle 1 Day 14: number analyzed (Participants) | 5 | 3
  Cycle 1 Day 14 | 138.0 (802.1) | 466.0 (104.7)

8. Secondary Outcome: Maximum Observed Concentration (Cmax) Of CC-486
Description: Maximum observed plasma concentration, obtained directly from the observed concentration versus time data.
Time Frame: as for outcome 6
Population: The PK population includes participants with evaluable CC-486 plasma PK profiles
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | CC-486 200 mg | CC-486 300 mg
Number analyzed (Participants) | 6 | 7
ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 4 | 6
  Cycle 1 Day 1 | 266.3 (53.8) | 170.7 (95.0)
  Cycle 1 Day 14: number analyzed (Participants) | 5 | 3
  Cycle 1 Day 14 | 102.7 (412.0) | 287.0 (50.7)

9. Secondary Outcome: Time to Reach Maximum Concentration (Tmax) Of CC-486
Description: Time to Cmax, obtained directly from the observed concentration versus time data.
Time Frame: as for outcome 6
Population: The PK population includes participants with evaluable CC-486 plasma PK profiles.
Measure: Median (Full Range); unit: Hours
Arm/Group | CC-486 200 mg | CC-486 300 mg
Number analyzed (Participants) | 6 | 7
Hours
  Cycle 1 Day 1: number analyzed (Participants) | 4 | 6
  Cycle 1 Day 1 | 1.0 [0.50 to 1.5] | 1.3 [0.50 to 1.5]
  Cycle 1 Day 14: number analyzed (Participants) | 5 | 3
  Cycle 1 Day 14 | 1.0 [0.0 to 2.0] | 1.0 [0.50 to 3.0]

10. Secondary Outcome: Terminal Half-Life (t1/2) of CC-486
Description: Terminal phase half-life in plasma, calculated as [(ln 2)/λz]. t1/2 was only calculated when a reliable estimate for λz could be obtained.
Time Frame: as for outcome 6
Population: The PK population includes participants with evaluable CC-486 plasma PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | CC-486 200 mg | CC-486 300 mg
Number analyzed (Participants) | 6 | 7
Hours
  Cycle 1 Day 1: number analyzed (Participants) | 4 | 6
  Cycle 1 Day 1 | 0.562 (23.1) | 0.635 (24.2)
  Cycle 1 Day 14: number analyzed (Participants) | 5 | 3
  Cycle 1 Day 14 | 0.584 (17.2) | 0.640 (32.0)

11. Secondary Outcome: Apparent Total Clearance (CL/F) Of CC-486
Description: Apparent volume of distribution, calculated as [(CL/F)/λz].
Time Frame: as for outcome 6
Population: The PK population includes participants with evaluable CC-486 plasma PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters/hour
Arm/Group | CC-486 200 mg | CC-486 300 mg
Number analyzed (Participants) | 6 | 7
Liters/hour
  Cycle 1 Day 1: number analyzed (Participants) | 4 | 6
  Cycle 1 Day 1 | 509.5 (58.3) | 845.3 (87.1)
  Cycle 1 Day 14: number analyzed (Participants) | 5 | 3
  Cycle 1 Day 14 | 1450 (802.1) | 643.7 (104.7)

12. Secondary Outcome: Apparent Volume of Distribution (Vz/F) Of CC-486
Description: Apparent volume of distribution, calculated as [(CL/F)/λz].
Time Frame: as for outcome 6
Population: The PK population includes participants with evaluable CC-486 plasma PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | CC-486 200 mg | CC-486 300 mg
Number analyzed (Participants) | 6 | 7
Liters
  Cycle 1 Day 1: number analyzed (Participants) | 4 | 6
  Cycle 1 Day 1 | 412.9 (42.9) | 774.6 (78.6)
  Cycle 1 Day 14: number analyzed (Participants) | 5 | 3
  Cycle 1 Day 14 | 1221 (581.3) | 594.8 (69.7)

ADVERSE EVENTS:
Time Frame: From Day 1 of study treatment until 28 days after the last dose of IP and those SAEs made known to the Investigator at any time thereafter that are suspected of being related to IP; up to final cut-off date of 08 August 2017; median duration of study treatment was 257 days for CC-486 200 mg and 114.5 days for CC-486 300 mg.
Arm/Group | CC-486 200 mg | CC-486 300 mg
All-Cause Mortality (participants affected / at risk) | 4/6 | 18/30
Serious Adverse Events (participants affected / at risk) | 4/6 | 12/30
Other Adverse Events (participants affected / at risk) | 6/6 | 29/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CC-486 200 mg (N=6) | CC-486 300 mg (N=30)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Asthenia (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 1
Pneumonia (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 1 | 0
Neutrophil count decreased (Investigations) | 2 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Brain oedema (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CC-486 200 mg (N=6) | CC-486 300 mg (N=30)
Anaemia (Blood and lymphatic system disorders) | 1 | 5
Leukopenia (Blood and lymphatic system disorders) | 0 | 4
Neutropenia (Blood and lymphatic system disorders) | 3 | 9
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 3
Sinus tachycardia (Cardiac disorders) | 1 | 0
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 2
Diabetes insipidus (Endocrine disorders) | 1 | 0
Eye oedema (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 3
Constipation (Gastrointestinal disorders) | 1 | 10
Dental caries (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 10
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 4
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 6 | 18
Oesophagitis (Gastrointestinal disorders) | 0 | 2
Stomatitis (Gastrointestinal disorders) | 2 | 4
Toothache (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 23
Asthenia (General disorders) | 0 | 8
Face oedema (General disorders) | 0 | 2
Facial pain (General disorders) | 0 | 2
Fatigue (General disorders) | 3 | 5
Hypothermia (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 2
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 8
Bacteraemia (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 1 | 1
Nasopharyngitis (Infections and infestations) | 0 | 2
Nosocomial infection (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 1 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 2
Skin infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 5
Aspartate aminotransferase increased (Investigations) | 1 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 2
Blood creatinine increased (Investigations) | 1 | 1
C-reactive protein increased (Investigations) | 0 | 2
Neutrophil count decreased (Investigations) | 1 | 1
Weight decreased (Investigations) | 0 | 5
Decreased appetite (Metabolism and nutrition disorders) | 2 | 8
Hyperammonaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 3
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Dizziness (Nervous system disorders) | 1 | 3
Dysgeusia (Nervous system disorders) | 0 | 2
Facial paralysis (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 1 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 2
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 3
Insomnia (Psychiatric disorders) | 1 | 2
Menstrual disorder (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 6
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The review of the efficacy data from the trial participants did not support proceeding to Stage 2 as the protocol-defined criteria of > 4 responders (a best response of CR or PR) in Stage 1 was not reached and study enrollment was stopped.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is more than 1 year from study completion. Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to 90 additional days. Investigator must delete confidential information before submission or defer publication to permit patent applications.

DOCUMENTS (5):
  • Study Protocol: CC-486-NPC-001_original protocol_Redacted.11July2014 (2014-07-11): https://cdn.clinicaltrials.gov/large-docs/43/NCT02269943/Prot_000.pdf
  • Study Protocol: CC-486-NPC-001.01.protocolAM1_RedactedOctober2014 (2014-10-01): https://cdn.clinicaltrials.gov/large-docs/43/NCT02269943/Prot_001.pdf
  • Study Protocol: CC-486-NPC-001_protocolAM2_Redacted.03April2015 (2015-04-03): https://cdn.clinicaltrials.gov/large-docs/43/NCT02269943/Prot_002.pdf
  • Study Protocol: CC-486-NPC-001_protocolAM3_Redacted.23September2016 (2016-09-23): https://cdn.clinicaltrials.gov/large-docs/43/NCT02269943/Prot_003.pdf
  • Statistical Analysis Plan (2017-05-15): https://cdn.clinicaltrials.gov/large-docs/43/NCT02269943/SAP_004.pdf